CLINICAL TRIAL: NCT03812523
Title: A Randomized Phase II Study Comparing Lorcaserin Versus Duloxetine for the Treatment of Chemotherapy-Induced Peripheral Neuropathy Produced by Oxaliplatin
Brief Title: Comparing Lorcaserin Versus Duloxetine for the Treatment of Chemotherapy-Induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeastern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA2018005 LVD
Record Dates: First submitted 2019-01-04; First posted 2019-01-23 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy
MeSH Terms: interventions — Duloxetine Hydrochloride; lorcaserin

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized controlled clinical trial in cancer patients receiving oxaliplatin treatment reporting neurotoxicity Grade 2 or higher by CTCAE guidelines to a member of their medical team. Enrollment goal is 50 patients. (25 evaluable patients per arm)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Coded Bottles
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Duloxetine 60 mg qd
  Interventions: Drug: Duloxetine 60 mg qd
- Intervention (Experimental): Lorcaserin 10 mg bid
  Interventions: Drug: Lorcaserin

INTERVENTIONS:
Drug: Duloxetine 60 mg qd — 60 mg tablet Taken by mouth, Once Daily for 180 Days
  Arms: Control
Drug: Lorcaserin — 10 mg tablet Taken by mouth Twice Daily for 180 Days
  Arms: Intervention

SUMMARY:
A Randomized Phase II study Comparing Lorcaserin versus Duloxetine for the Treatment of Chemotherapy-Induced Peripheral Neuropathy Produced by Oxaliplatin

DETAILED DESCRIPTION:
To examine lorcaserin a selective R-HT2c receptor antagonist approved by FDA as weight loss drug- for its ability to improve proprioceptive movements in patients with advanced colorectal cancer who developed neurotoxicity during oxaliplatin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of invasive colorectal cancer, locally advanced or advanced, requiring oxaliplatin-based chemotherapy for treatment.
* Subject has agreed to receive treatment at Cancer Treatment Centers of America, Southeastern Regional Medical Center.
* Subject is Male or Female
* Subject is 18 years of age or older.
* Subject is a patient who reports neurotoxicity symptom grade 2 or more according CTCAE criteria to his or her medical oncologist following one or more cycles of oxaliplatin-based chemotherapy treatment.
* Subject is a patient who is capable and accepting of completing study questionnaires at each data collection point.
* Subject has adequate English fluency for completion of data collection. The surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.
* Subject must have the ability to understand and the willingness to sign a written informed consent
* Subject must be willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Subjects who have previously been exposed to neurotoxic agents including pyridoxine (>100 mg/day), colchicine, allopurinol, or phenytoin;
* Subjects with pre-existing comorbidities, such as: diabetes, uremia, significant peripheral vascular disease, HIV, or progressive or degenerative neurologic disorders (e.g., multiple sclerosis, B12 deficiency); cardiovascular valve disease, history of cardiovascular event,
* Subjects with a history of lumbosacral laminectomy or radiculopathy;
* Subjects who have been prescribed and taken gabapentin, pregabalin, or duloxetine currently or within the last 1 months)
* Subjects who have established or suspected family history of inherited neuropathy.
* Subjects unable to swallow indicated medication
* Subjects in general with a medical condition, laboratory finding, or physical exam finding that precludes participation
* Subject weight of ≥350 lbs.
* Subjects who currently use disallowed concomitant medications
* Subjects with any form of cardiac implants
* Subjects who report recent febrile illness that precludes or delays participation
* Subjects with pregnancy or lactation
* Subjects with known allergic reactions to components of the study product(s)
* Subjects receiving treatment with another investigational drug or other intervention
* Subjects with a history of or current tobacco or illegal substance use
* Subjects exhibiting significant psychiatric or cognitive impairment (dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Assessment with respect to duloxetine of the effect of lorcaserin on the Pain Numerical Rating Scale. | 180 days
  Duloxetine efficacy as Measured by Pain Score 0-10 Numerical Rating Scale. Subject will rate level of pain experienced from 0 (No Pain) to 10 (Worst Possible Pain) for each question on the Brief Pain Inventory Short Form. A rating of 5 would be Moderate Pain.
Assessment with respect to duloxetine of the effect of lorcaserin on the patient-reported quality of life. | 180 days
  Subject quality of life will be measured using the Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group-Neurotoxocity (FACT/GOG-NTX) Questionnaire. For each statement, the subject will answer 0-5 with 0 being "Not at All" and 5 being "Very Much"
Assessment with respect to duloxetine of the effect of lorcaserin on the patient-reported quality of life. | 180 days
  Subject quality of life will also be measured using the MD Anderson Symptom Inventory (MDASI) Questionnaire, with CTCA addendum. For each statement, the subject will answer from 0-10, with 0 being "Not Present" and 10 being "As Bad as You Can Imagine)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Treatment Centers of America - Atlanta, Newnan, Georgia, United States